CLINICAL TRIAL: NCT06218914
Title: Open-label, Phase 1, Multi-Center Master Protocol to Evaluate the Safety and Preliminary Anti-Tumor Activity of TCR-engineered T Cells Recognizing KRAS Mutations in Adult Subjects With Unresectable, Advanced, and/or Metastatic Solid Tumors
Brief Title: Phase 1 Study to Investigate TCRTs KRAS Mutation in Unresectable, Advanced, and/or Metastatic Solid Tumors
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: NT-112-301
Record Dates: First submitted 2024-01-09; First posted 2024-01-23 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: Non-small Cell Lung Cancer; Colorectal Carcinoma; Pancreatic Ductal Adenocarcinoma; Endometrial Cancer; Solid Tumor, Adult; KRAS G12D
Keywords: TCR-T cell therapy; KRAS; KRAS G12D; Autologous; PDAC; NSCLC; Colorectal Cancer; Solid tumors; Pancreatic Ductal Adenocarcinoma; HLA-C*08:02; HLA-A*11:01; HLA-A*11:02
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Colorectal Neoplasms; Endometrial Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- NT-112 (Experimental): Part A Dose Escalation and Part B Dose Expansion of NT-112
  Interventions: Biological: NT-112: Autologous, engineered T Cells targeting KRAS G12D
- AZD0240 (Experimental): Part A Dose Escalation and Part B Dose Expansion of AZD0240
  Interventions: Biological: AZD0240: Autologous, engineered T Cells targeting KRAS G12D

INTERVENTIONS:
Biological: NT-112: Autologous, engineered T Cells targeting KRAS G12D — NT-112 targets KRAS G12D in the context of HLA-C*08:02
  Arms: NT-112
Biological: AZD0240: Autologous, engineered T Cells targeting KRAS G12D — AZD0240 targets KRAS G12D in the context of HLA-A*11:01 or HLA-A*11:02
  Arms: AZD0240

SUMMARY:
Phase I Study, a master protocol to investigate TCR-Engineered T cells recognizing KRAS mutations in adult subjects with Unresectable, Advanced, and/or Metastatic Solid Tumors.

DETAILED DESCRIPTION:
This is a Phase 1, open-label, Phase 1, Multi-Center Master Protocol to evaluate the safety and preliminary Anti-Tumor activity of TCR-Engineered T cells (KRAS TCRTs) recognizing KRAS mutations in adult subjects with Unresectable, Advanced, and/or Metastatic Solid Tumors.

ELIGIBILITY:
Key Inclusion Criteria:

* Age ≥18 years
* Diagnosed with NSCLC, Colorectal adenocarcinoma, Pancreatic adenocarcinoma, Endometrial Cancer or any other solid tumor
* Tumors must harbor a KRAS G12D variant mutation and subject must be HLA-C*08:02 positive, HLA-A*11:01 or HLA-A*11:02 positive in at least one allele
* Subject has advanced solid cancer, defined as unresectable, advanced, and/or metastatic disease (Stage III or IV) after at least 1 line of approved systemic standard of care (SOC) treatment regimen and for which there are no available curative treatment options.
* Presence of at least 1 measurable lesion per RECIST v1.1
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 1 at the time of enrollment

Key Exclusion Criteria:

* Any other primary malignancy within the 3 years prior to enrollment (except for non-melanoma skin cancer, carcinoma in situ (eg, cervix, bladder, breast) or low-grade prostate cancer
* Known, active primary central nervous system (CNS) malignancy
* History of prior adoptive cell and gene therapy, allogeneic stem cell transplant or solid organ transplantation.
* History of stroke or transient ischemic attack within the 12 months prior to enrollment.
* History of clinically significant cardiac disease within the 6 months prior to enrollment or heart failure at any time prior to enrollment.
* Systemic therapy within at least 2 weeks or 3 half-lives, whichever is shorter, prior to enrollment.
* Any form of primary immunodeficiency.
* Active immune-mediated disease requiring systemic steroids or other immunosuppressive treatment (except if related to prior checkpoint inhibitor therapy)
* Female of childbearing potential who is lactating or breast feeding at the time of enrollment
* Prior treatment with pan-KRAS or KRAS G12D targeting agents unless presence of KRAS G12D mutation is confirmed after the completion of treatment with pan-KRAS or KRAS G12D targeting agents.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2024-03-22 (Actual); Primary Completion 2027-08-30 (Estimated); Study Completion 2043-11-18 (Estimated)

PRIMARY OUTCOMES:
Part A (Dose Escalation): Evaluate the safety of KRAS TCRTs in subjects with unresectable, advanced, and/or metastatic solid tumors | Through study completion, an average of 2 years
  Incidence of DLTs, treatment-emergent adverse events (TEAEs) and serious adverse events (SAEs)
Part A (Dose Escalation): Evaluate MTD and recommended dose for expansion (RDE) | 28 days after infusion
  Incidence of DLTs, treatment-emergent adverse events (TEAEs) and serious adverse events (SAEs)
Part B (Expansion): Further evaluate the safety of KRAS TCRTs at the RDE in subjects with unresectable, advanced, and/or metastatic solid tumors | 28 days after infusion
  Incidence of DLTs, treatment-emergent adverse events (TEAEs), and serious adverse events (SAEs)

SECONDARY OUTCOMES:
Part A (Dose Escalation): Evaluate the preliminary anti-tumor activity of KRAS TCRTs in subjects with unresectable, advanced, and/or metastatic solid tumors | Up to 24 months post-infusion
  Objective response rate (ORR) per Response Evaluation Criteria in Solid Tumors (RECIST) v1.1, determined by Investigator assessment
  * Best objective response (BOR)
  * Duration of response (DOR)
  * Clinical benefit rate (CBR) (complete response [CR], partial response [PR], stable disease [SD])
  * Time to response (TTR)
  * Progression-free survival (PFS)
  * Overall survival (OS)
Part B (Dose Expansion): Evaluate the preliminary anti-tumor activity of KRAS TCRTs at the RDE in subjects with unresectable, advanced, and/or metastatic solid tumors | Up to 24 months post infusion
  Objective response rate (ORR) per Response Evaluation Criteria in Solid Tumors (RECIST) v1.1, determined by Investigator assessment
  * Best objective response (BOR)
  * Duration of response (DOR)
  * Clinical benefit rate (CBR) (complete response [CR], partial response [PR], stable disease [SD])
  * Time to response (TTR)
  * Progression-free survival (PFS)
  * Overall survival (OS)

CONTACTS AND LOCATIONS:
Locations (16):
- United States (16):
  - Research Site, Duarte, California
  - Research Site, Los Angeles, California
  - Research Site, Newport Beach, California
  - Research Site, Jacksonville, Florida
  - Research Site, Chicago, Illinois
  - Research Site, Westwood, Kansas
  - Research Site, St Louis, Missouri
  - Research Site, New York, New York
  - Research Site, Philadelphia, Pennsylvania
  - Research Site, Pittsburgh, Pennsylvania
  - Research Site, Nashville, Tennessee
  - Research Site, Dallas, Texas
  - Research Site, Galveston, Texas
  - Research Site, Houston, Texas
  - Research Site, Aberdeen, Washington
  - Research Site, Milwaukee, Wisconsin

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal Vivli.org. All requests will be evaluated as per the AZ disclosure commitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure
  Yes, indicates that AZ are accepting requests for IPD, but this does not mean all requests will be shared.
Supporting Information: Study Protocol, SAP
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA PhRMA Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the anonymized individual patient-level data via secure research environment Vivli.org. Signed Data Usage Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information.
URL: https://vivli.org/